CLINICAL TRIAL: NCT05559944
Title: Brief Writing Programs for Sexual Minority Young Adults in Alabama
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study never started as changes to the study structure were determined by the community advisory board overseeing the project prior to study start.
Sponsor: Auburn University (Other)
Responsible Party: Principal Investigator, Tiffany Brown, Assistant Professor, Auburn University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: #22-317
Record Dates: First submitted 2022-09-19; First posted 2022-09-29 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Expressive Writing; Self-Affirmation; Control
Keywords: LGBTQIA+; Body Image; Alabama; Eating Disorders
MeSH Terms: conditions — Feeding and Eating Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Expressive Writing (Experimental): Participants will be asked to write about the biggest body image or eating-related stressor they have experienced as a member of the LGBTQ+ community. A general list of the types of stressors and contexts commonly described will be provided to participants, given that meta-analytic research supports that providing examples enhances the efficacy of expressive writing.
  Interventions: Behavioral: Expressive Writing
- Self-Affirmation (Experimental): Participants will respond to one new vignette per day describing a SM young adult experiencing severe body image stress in Alabama. Participants will be asked to write to this person and provide advice based on their own experience as a SM young adult. Vignettes will be identical across participants; however, they will be matched to participants' sexual identity, gender identity, and race/ethnicity.
  Interventions: Behavioral: Self-Affirmation
- Control (Placebo Comparator): Consistent with prior research participants will write about their routine daily activities since waking up for 20 minutes each day, sans emotional content.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Expressive Writing — Participants will be asked to write about the biggest body image or eating-related stressor they have experienced as a member of the LGBTQ+ community.
  Arms: Expressive Writing
Behavioral: Self-Affirmation — Participants will receive one new vignette per day describing a SM young adult experiencing severe body image stress in Alabama. Participants will be asked to write to this person and provide advice based on their own experience as a SM young adult. Vignettes will be identical across participants; however, they will be matched to participants' sexual identity, gender identity, and race/ethnicity.
  Arms: Self-Affirmation
Behavioral: Control — Consistent with prior research participants will write about their routine daily activities since waking up for 20 minutes each day, sans emotional content.
  Arms: Control

SUMMARY:
Sexual minority (SM; e.g., gay, lesbian, bisexual, pansexual, queer) young adults are at elevated risk for eating disorders (EDs). Researchers have used minority stress theory to understand how increased risk is due, in part, to stigma and discrimination from being part of a marginalized group. Despite this glaring inequity, limited programs exist to prevent EDs in SM populations. Critically, many SM young people live in rural regions with high anti-LGBTQ+ stigma and limited access to SM-specific resources. The proposed project will address this gap by adapting and evaluating two brief online interventions to reduce ED risk. N = 120 SM young adults in rural regions of Alabama with high LGBTQ+ stigma and low SM-specific resources will be randomized into one three brief online writing interventions: 1) expressive writing (n = 40), 2) self-affirmation (n = 40), or 3) control (n = 40). Participants will complete assessments pre-intervention, post-intervention, and 1-month post-intervention. Aim 1 will assess intervention feasibility and acceptability. Aim 2 will compare the brief online writing interventions to control in improving body image and ED symptoms. Finally, an exploratory aim will examine posited intervention mechanisms and whether the level of SM stigma and discrimination participants experience pre-intervention impacts intervention efficacy. This research will help support and benefit underserved SM young adults by filling a critical need for brief, scalable interventions that can be delivered online to help reduce ED risk. Data from this project will serve as pilot data for a subsequent R-series grant application from NIH.

ELIGIBILITY:
Inclusion Criteria:

* ages 18-30
* identify as SM (gay, lesbian, bisexual, pansexual, or queer)
* endorse body dissatisfaction
* currently living in one of the following AL counties: Lee, Dallas, Lowndes, Autauga, Coosa, Elmore, Tallapoosa, Macon, or Russell
* have internet access (either via computer/tablet, mobile phone, or community center[e.g., library])

Exclusion Criteria:

* meet criteria for an ED, based on self-report screener
* non-English speaking
* Lack of internet access
* Not living in one of the following AL counties: Lee, Dallas, Lowndes, Autauga, Coosa, Elmore, Tallapoosa, Macon, or Russell
* Younger than 18, older than 30

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2024-12 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Body Image | changes from baseline through 1-month follow-up
  Body Image States Scale (BISS); 7-item self-report measure about satisfaction with overall appearance. Scores range from 1-9, with higher scores reflecting more positive body image
Eating Disorder Symptoms | changes from baseline through 1-month follow-up
  Eating Pathology Symptom Inventory (EPSI); 45-item measure that assesses 8 domains of eating disorder pathology, scores range from 0-32, with higher scores indicating greater pathology

SECONDARY OUTCOMES:
Internalization of Appearance Ideals and Pressures | changes from baseline through 1-month follow-up
  Sociocultural Attitudes Towards Appearance Scale-4 (SATAQ-4); 22-item measure of internalization of appearance ideals and pressures. Scores range from 4-25, with higher scores indicating greater appearance internalization
Negative Affect | changes from baseline through 1-month follow-up
  Depression, Anxiety, and Stress Scale (DASS-21); 21 item measure used to assess depression, anxiety, and nonspecific physiological arousal which load onto a higher order factor of psychological distress/negative affect. Scores range from 0-63, with higher scores indicating greater negative affect
Interpersonal Emotion Regulation | changes from baseline through 1-month follow-up
  Difficulties in Interpersonal Regulation of Emotion (DIRE); 24-item measures of maladaptive interpersonal emotional regulation. Scores range from 3-30 and higher scores indicate greater pathology.
Health-related quality of life | changes from baseline through 1-month follow-up
  World Health Organization Quality of Life- (WHO-BREF); 26-item self-report measure for physical and psychological social relationships and environmental health. Scores range from 4-20; higher scores indicate a better quality of life.
Social Self-Esteem | changes from baseline through 1-month follow-up
  Social Self-Esteem Scale (SSES); Measures confidence and self-esteem in social situations across 9 items. Scores range from 9-54, with higher scores indicating grater social self-esteem.
Self-Stigma of Seeking Help | changes from baseline through 1-month follow-up
  Self-Stigma of Seeking Help (SSOSH); Stigma surrounding seeking help for psychological concerns. Scores range from 10-50, with higher scores indicating greater stigma.
Substance Use | changes from baseline through 1-month follow-up
  Alcohol, Smoking, and Substance Involvement Screening (ASSIST); Examines alcohol and substance use patterns. Scores range from 0-39 and higher scores reflect greater substance use problems.

OTHER OUTCOMES:
Coping Self-Efficacy | Baseline
  Coping Self Efficacy Scale (CSES); Assesses sexual minority(SM)-stress coping self efficacy, as adapted for address SM stress in prior research (13 items, 11-point scale, range 0-130, higher scores indicate greater SM-stress coping self-efficacy).
Discrimination | Baseline
  Heterosexist Harassment, Rejection, and Discrimination Scale; Measure assesses experiences with victimization and rejection related to SGM identity (14 items, scores range from 14-84, with higher scores reflecting greater experiences with discrimination)
Internalized Stigma | Baseline
  Internalized Homophobia Scale (IHP); Assess internalization of negative attitudes toward one's sexual identity (9 items, scores range from 5-45, higher scores indicate greater internalized stigma)
Sexual Orientation Concealment | Baseline
  Sexual Orientation Concealment Scale (SOCS); Assess the degree to which one intentionally conceals their sexual identity (6 items, scores range from 6-30, higher scores indicate greater concealment)
Rejection Sensitivity | Baseline
  Sexual Minority Women (or Gay-Related) Rejection Sensitivity; Assesses sensitivity towards rejection due to sexual identity (14-16 items, ranges 1-36, higher scores indicate greater rejection sensitivity)
Community Involvement | Baseline
  Items from the Social Justice Sexuality Survey include 6 items of LGBTQ community involvement (range 6-36, higher scores indicate greater community involvement)
Intraminority Stress | Baseline
  Abbreviated Intraminority Stress Scale; Assesses stressors within the gay community (8 items, range 8-40, higher scores indicate greater perception of community stress)

CONTACTS AND LOCATIONS:
Overall Officials: Jordan Merriweather, Study Director — Auburn University

IPD SHARING:
Plan to Share IPD: No
Data will be maintained for 5 years following the close of the study. Those interested in learning more about the data can contact the Principal Investigator (tab0110@auburn.edu)

REFERENCES:
- See also: Contact Page for Study Enrollment and Information — https://acceptlab.wixsite.com/acceptlab/contact